CLINICAL TRIAL: NCT00363337
Title: A Preliminary Study of the Effectiveness and Tolerability of Aripiprazole in Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Susan McElroy, Lindner Center of HOPE
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-Parker
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Bipolar Depression
Keywords: Adults; Bipolar Depression; Bipolar Disorder; Bipolar I; Bipolar II; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Aripiprazole

INTERVENTIONS:
Drug: aripiprazole — open label treatment with aripiprazole
  Other Names: Abilify

SUMMARY:
The specific aim of this study is to obtain preliminary evidence of the acute effectiveness and tolerability of aripiprazole in the treatment of bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* subjects must have bipolar I, II or NOS disorder as defined by DSM-IV-TR; must have clinical significant depressive symptoms and have failed one or more mood stabilizer trials; may or may not be receiving antimanic or mood stabilizing medications; subjects or legally authorized representative must sign the Informed Consent document after the nature of the trial has been fully explained; if female, subjects must be postmenopausal, surgically incapable of childbearing or practicing medically acceptable effective method(s) of contraception.

Exclusion Criteria:

* subjects who do not have bipolar disorder by DSM-IV criteria; subjects with current DSM-IV Axis I diagnosis of delirium, dementia, amnesia or other cognitive disorders or a psychotic disorder; subjects with serious general medical illness; subjects who are allergic to or have demonstrated hypersensitivity to aripiprazole; women who are pregnant or nursing; subjects who have received an experimental drug or used an experimental device within 30 days; subjects who have a history of neurologic malignant syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | per protocol

SECONDARY OUTCOMES:
Clinical Global Impression Scale Modified for Bipolar Illness (CGI-BP) | per protocol

CONTACTS AND LOCATIONS:
Overall Officials: Susan L McElroy, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] McElroy SL, Suppes T, Frye MA, Altshuler LL, Stanford K, Martens B, Leverich GS, Post RM, Keck PE Jr. Open-label aripiprazole in the treatment of acute bipolar depression: a prospective pilot trial. J Affect Disord. 2007 Aug;101(1-3):275-81. doi: 10.1016/j.jad.2006.11.025. Epub 2007 Jan 16. PMID 17229469